CLINICAL TRIAL: NCT06946953
Title: Translational Application of Airway Basal Stem Cell Therapy in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Airway Basal Stem Cell Therapy in Chronic Obstructive Pulmonary Disease (COPD)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250322
Record Dates: First submitted 2025-03-22; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients (Experimental)
  Interventions: Biological: P63+ lung progenitors

INTERVENTIONS:
Biological: P63+ lung progenitors — 1. Patient Screening and Cell Collection:
     Eligible patients will undergo sample collection at the study center or authorized tertiary hospitals. The operator will collect samples via bronchial brushing from three healthy segments of the patient's 3-5 level bronchi. The samples will be transported to a cooperative production facility for isolation and preparation. The cell preparation cycle is approximately 4-8 weeks. Patients will bear the costs of this process.
  2. Transplantation Therapy:
     Transplantation therapy will be conducted at Ruijin Hainan Hospital. The cell preparation will be administered via fiberoptic bronchoscopy to each lung segment, with one dose per patient. After infusion, patients are advised to remain hospitalized for 24-48 hours for observation.
  3. Post-Treatment Follow-Up:
  Patients are advised to return for examination and evaluation at 4 and 24 weeks post-treatment.
  Other Names: Lung progenitors; Airway basal stem cells

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of REGEND001, an autologous bronchial basal cell therapy, for the treatment of Chronic Obstructive Pulmonary Disease (COPD). COPD is a chronic respiratory condition characterized by persistent airflow limitation and impaired lung function, leading to significant morbidity and mortality worldwide. Current treatments primarily focus on symptom management and have limited impact on disease progression or survival. This study proposes a novel approach using autologous bronchial basal cells, which have demonstrated the potential to repair damaged lung tissue and improve lung function in preclinical studies. The therapy involves the collection of bronchial basal cells via bronchial brushing, followed by their expansion and reintroduction into the patient's lungs via bronchoscopic infusion. The primary objective is to assess the improvement in lung diffusion capacity (DLCO), with secondary endpoints including changes in lung ventilation function (FEV1, FVC) and quality of life (CAT score). The study will also monitor safety, including the incidence of adverse events. Eligible participants are COPD patients aged 40-80 with moderate to severe disease. The trial includes a screening phase, cell collection, transplantation, and follow-up assessments at 4 and 24 weeks post-treatment. This study represents a promising advancement in regenerative medicine for COPD, offering a potential therapeutic option that addresses the underlying structural damage in the lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with COPD according to the 2021 Global Initiative for Chronic Obstructive Lung Disease (GOLD);
2. Post-bronchodilator FEV1/FVC <70%;
3. DLCO ≥20% and <80% of predicted value.

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant within 1 year after treatment (or male participants planning for their spouse to become pregnant);
2. Positive for syphilis (TP-Ab), HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies;
3. Current or past history of malignancy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in DLCO from baseline. | Baseline, 4 weeks post treatment, 24 weeks post treatment
  The diffusing capacity of the lungs for carbon monoxide (DLCO) is a measurement of the gas transfer capacity of lung.

SECONDARY OUTCOMES:
Change in FEV1 from baseline. | Baseline, 4 weeks post treatment, 24 weeks post treatment
Change in FVC from baseline. | Baseline, 4 weeks post treatment, 24 weeks post treatment
Improvement in CAT score (symptoms, activity, and psychological status). | Baseline, 4 weeks post treatment, 24 weeks post treatment
  CAT, COPD Assessment Test. Score range: 0 to 40. Higher scores indicate a worse outcome.

OTHER OUTCOMES:
Incidence of adverse events and serious adverse events. | Through study completion, an average of 6 months
  Safety Evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China